CLINICAL TRIAL: NCT04413539
Title: Evaluation of Impact of Disease on Quality of Life, Education and Socio-professional Integration of Adults and Parents of Children Living with Sickle- Cell Disease in France
Acronym: DREPAtient
Status: Completed | Type: Observational
Sponsor: Argo Sante (Other)
Collaborators: Filière de santé maladies rares MCGRE (Unknown); Fédération des malades drépanocytaires et thalassémiques SOS Globi (Unknown); Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2020-A00729-30
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2021-07

CONDITIONS: Sickle-cell Disease (SCD)
Keywords: Sickle-cell disease; quality of life; education; socio-professional integration; france
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Sickle cell disease (SCD) is the most common genetic disease in France. Its consequences on patient's life-course and quality of life need to be precisely identified among French patients and their family to be able to improve patients care according to their specific needs.

The aim of the study is to accurately describe the impact of SCD on quality of life of patients living in France, or their family (for minor patients). The consequences of the disease on professional life, education and material condition of patients or their parents will be described by the patients themselves.

DETAILED DESCRIPTION:
This is a retrospective study. Patients or parents of minor patients living in France and suffering from SCD will be informed about the study and enrolled during their usual follow-up, or by patients' associations. They will be asked to answer an anonymous survey online relating to their whole life-course with SCD and exploring different aspects of the consequences of the disease on their life. It contains 4 different sections:

1. socio-demographic questions to establish a respondent profile
2. health status of the respondent to establish the severity of the disease
3. education, professional life, material and economic situation
4. quality of life through MOS SF-36 questionnaire This is a one-shot survey, which will take approximatively 20 to 30 minutes to answer by the respondent.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Diagnosed with SCD or parent of a minor child diagnosed with SCD
* Able to speak and understand French
* Willing to participate to the study

Exclusion Criteria:

* Person having serious difficulties to read or speak French, unable to answer the questions
* Person suffering from other chronic disease which could bias the representation they have about SCD
* Patient cured with a bone marrow transplant
* Patient with mental disorder preventing the patient to understand the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults or parents of minor children with SCD living in France.
Sampling Method: Non-Probability Sample
Enrollment: 1088 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2021-04-27 (Actual)

PRIMARY OUTCOMES:
Describe the disease impact on quality of life through description of professional life, education and material condition of patients, or their parents (for minor patients), suffering from sickle-cell disease and living in France. | Once at enrollment
  Measure of mutual impact of health status on patients educational and socio-professional life course.

SECONDARY OUTCOMES:
- Study the factors of heterogeneity of patients' profiles - Explore the causal relation between health status and employment conditions, education, material and economic situation - Assess the patients' needs in care and socio-economic support | Once at enrollment
  The perceived impact of disease on education will be confirmed by:
  * Type of education adjustment introduced
  * The level and the cause of leaving full-time education
  * The intensity of school absences
  * The feeling of discrimination on school time
  The impact of disease on professional life will be measured by:
  * The professional status
  * The sick leaves
  * The feeling of discrimination at work
  * The compatibility of work conditions with the disease
  The impact of disease on material and economic situation will be assessed by:
  * The income level
  * The patient cost sharing
  * The remaining balance
  * The recognition of handicap
  * The recognition of disability
  The quality of life score of respondents:
  - Medical outcome study short form 36 item health survey (MOS SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Frederic Galacteros, MD,PhD,Prof., Principal Investigator — Red Cell genetic diseases unity, Henri Mondor Hospital, Paris
Locations (1):
- Centre de références syndromes drépanocytaires majeurs thalassémie et autres maladies rares du globule rouge et de l'érythropoïése, Créteil, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Crosby LE, Joffe NE, Irwin MK, Strong H, Peugh J, Shook L, Kalinyak KA, Mitchell MJ. School Performance and Disease Interference in Adolescents with Sickle Cell Disease. Phys Disabil. 2015;34(1):14-30. doi: 10.14434/pders.v34i1.13918. PMID 27547816
- [Background] Dos Santos JP, Gomes Neto M. Sociodemographic aspects and quality of life of patients with sickle cell anemia. Rev Bras Hematol Hemoter. 2013;35(4):242-5. doi: 10.5581/1516-8484.20130093. PMID 24106440
- [Background] Gardner K, Douiri A, Drasar E, Allman M, Mwirigi A, Awogbade M, Thein SL. Survival in adults with sickle cell disease in a high-income setting. Blood. 2016 Sep 8;128(10):1436-8. doi: 10.1182/blood-2016-05-716910. Epub 2016 Jul 20. No abstract available. PMID 27439910
- [Background] Habibi A, Arlet JB, Stankovic K, Gellen-Dautremer J, Ribeil JA, Bartolucci P, Lionnet F; centre de reference maladies rares << syndromes drepanocytaires majeurs >>. [French guidelines for the management of adult sickle cell disease: 2015 update]. Rev Med Interne. 2015 May 11;36(5 Suppl 1):5S3-84. doi: 10.1016/S0248-8663(15)60002-9. French. PMID 26007619
- [Background] Chapelon E, Garabedian M, Brousse V, Souberbielle JC, Bresson JL, de Montalembert M. Osteopenia and vitamin D deficiency in children with sickle cell disease. Eur J Haematol. 2009 Dec 1;83(6):572-8. doi: 10.1111/j.1600-0609.2009.01333.x. Epub 2009 Aug 13. PMID 19682065
- [Background] Godeau B, Noel V, Habibi A, Schaeffer A, Bachir D, Galacteros F. [Sickle cell disease in adults: which emergency care by the internists?]. Rev Med Interne. 2001 May;22(5):440-51. doi: 10.1016/s0248-8663(01)00369-1. French. PMID 11402515
- [Background] LINDENBAUM J, KLIPSTEIN FA. FOLIC ACID DEFICIENCY IN SICKLE-CELL ANEMIA. N Engl J Med. 1963 Oct 24;269:875-82. doi: 10.1056/NEJM196310242691701. No abstract available. PMID 14050985
- [Background] Noll RB, Vannatta K, Koontz K, Kalinyak K, Bukowski WM, Davies WH. Peer relationships and emotional well-being of youngsters with sickle cell disease. Child Dev. 1996 Apr;67(2):423-36. doi: 10.1111/j.1467-8624.1996.tb01743.x. PMID 8625722
- [Background] Rees DC, Williams TN, Gladwin MT. Sickle-cell disease. Lancet. 2010 Dec 11;376(9757):2018-31. doi: 10.1016/S0140-6736(10)61029-X. Epub 2010 Dec 3. PMID 21131035
- [Background] Salih KMA. The impact of sickle cell anemia on the quality of life of sicklers at school age. J Family Med Prim Care. 2019 Feb;8(2):468-471. doi: 10.4103/jfmpc.jfmpc_444_18. PMID 30984656
- [Background] Sehlo MG, Kamfar HZ. Depression and quality of life in children with sickle cell disease: the effect of social support. BMC Psychiatry. 2015 Apr 11;15:78. doi: 10.1186/s12888-015-0461-6. PMID 25880537
- See also: Related Info — https://www.modalisa-enquete.com/drepatient